CLINICAL TRIAL: NCT03090711
Title: Sleep as a Model to Understand and Manipulate Cortical Activity in Order to Promote Neuroplasticity and Functional Recovery After Stroke
Brief Title: Sleep as a Model to Understand and Manipulate Cortical Activity in Order to Promote Functional Recovery After Stroke
Acronym: SSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2016-01387
Record Dates: First submitted 2017-03-09; First posted 2017-03-27 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Hemispatial Neglect
MeSH Terms: conditions — Perceptual Disorders | interventions — Transcranial Magnetic Stimulation; Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TMS (Experimental): Real transcranial magnetic stimulation (TMS).
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- sham TMS (Sham Comparator): Sham transcranial magnetic stimulation (TMS) as a comparison.
  Interventions: Device: sham Transcranial Magnetic Stimulation (TMS)
- TMS and tACS (Experimental): Real transcranial magnetic stimulation (TMS) and real transcranial alternating current stimulation (tACS).
  Interventions: Device: Transcranial Magnetic Stimulation (TMS); Device: Transcranial Alternating Current Stimulation (tACS)
- TMS and sham tACS (Sham Comparator): Real transcranial magnetic stimulation (TMS) and sham transcranial alternating current stimulation (tACS) as a comparison.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS); Device: sham Transcranial Alternating Current Stimulation (tACS)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — The investigators recently showed that the repeated application of the so-called continuous theta burst protocol (cTBS) over the contralesional hemisphere resulted in a long-standing improvement of visual hemineglect (Cazzoli et al., 2012). The cTBS protocol was developed by Huang et al. (Huang et al., 2005) and modified by the investigators' group (Nyffeler et al., 2006). TBS protocol consists of a burst of 3 pulses at a frequency of 30 Hz, repeated at 6 Hz. One continuous train includes 801 pulses, the duration of one cTBS train is 44 seconds.
  Arms: TMS; TMS and sham tACS; TMS and tACS
Device: Transcranial Alternating Current Stimulation (tACS) — TACS stimulation involves two electrodes placed on either side of the desired site of cortical stimulation. The mode of stimulation used in this experiment is identical to previous studies using tACS in sleep ( Marshall et al., 2006; Prehn-Kristensen et al., 2014 ). Stimulation follows a sinusoidal pattern from 0 to 260 μA. This pattern is delivered at 0.75 Hz and is repeated for 225 cycles; a total of 5 minutes of stimulation. This 5 minute pattern is again repeated 5 times, with a minute of no stimulation between each; thus for a total of 30 minutes.
  Arms: TMS and tACS
Device: sham Transcranial Magnetic Stimulation (TMS) — Sham coil will be used to exclude possible nonspecific effects of the TMS. The sham coil is shielded i.e., the magnetic field output is weakened and therefore insufficiently powerful to stimulate the cortex.
  Arms: sham TMS
Device: sham Transcranial Alternating Current Stimulation (tACS) — Sham stimulation will be used to exclude possible nonspecific effects of the tACS. Sham tACS stimulation will involve actual stimulation for the first 30 seconds of the ramp-up period (stimulation power is gradually increased until its final level), and then immediately gradually decreased until zero (without the intermediate 4 minutes of actual stimulation). This procedure will be repeated 5 times every 6 minutes and shall induce similar cutaneous sensations as real stimulation.
  Arms: TMS and sham tACS

SUMMARY:
Brain functions are supported by multiple cell types, including neuronal and non-neuronal cells that are connected into complex networks. When the connectivity between those cells is altered or disrupted, the functioning of the brain is impaired. In stroke, the interruption of blood supply to the neural circuits results in connectivity damage and permanent disabilities. Experimental evidence suggests that some types of brain state, including sleep, can protect brain tissue from stroke and "repair" the damaged circuits. This project will investigate the neuronal mechanism underlying the protective effect of sleep on brain connectivity and network activity. To this end, the investigators will use a collection of state-of-the-art technologies including high-density electroencephalography (hd-EEG), transcranial magnetic stimulation (TMS) and transcranial alternating current stimulation (tACS). Perspectives include a better understanding of the causes and consequences of the perturbed electrical activity of the brain during sleep in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature
* Age between 18 and 80 years
* First-ever right-sided stroke
* Normal or corrected to normal vision
* Demonstration of left hemispatial neglect (after a right-hemispheric brain lesion) found in a comprehensive neuropsychological test battery and clinical assessment
* At least 3 weeks post-stroke

Exclusion Criteria:

* Concomitant neurodegenerative diseases
* Psychiatric diseases
* Decompressive craniectomy
* History of documented sleep disorders in the medical record (e.g. insomnia, hypersomnia, rem-sleep behaviour disorder)
* Epileptic seizures
* Implanted medical devices (e.g.: pacemakers, cochlear implants, implanted neurostimulators)
* Presence of metal in the region of the head (excluding fixed dental implants such as tooth fillings or fixed dental braces)
* Medication with drugs possibly lowering the seizure threshold
* Alcohol or drug abuse
* Inability to follow the procedures of the study
* For female patients: in order to participate in the study, female patients in reproductive age need to take a pregnancy test (a standard urine pregnancy test will be provided).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in visual exploration and sleep parameters and the effect of cTBS | Day 3
  Relationship of visual exploration (mean cumulative fixation duration) to sleep parameters (slow wave activity and spindles) from the baseline to post-cTBS sleep.
Change from baseline in the effect of tACS on visual exploration | Day 2
  Group comparison of visual exploration task (mean cumulative fixation duration) between real and sham tACS.

SECONDARY OUTCOMES:
The effect of cTBS on sleep | Day 1 to 3
  Relationship between baseline sleep parameters (slow wave activity and spindles) and effectiveness of cTBS.
The effect of tACS on sleep | Day 1 to 2
  Change in sleep architecture (REM and NREM sleep) between tACS and sham stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio L. Bassetti, Prof. Dr. med., Principal Investigator — Department of Neurology, Inselspital, Bern University Hospital
Locations (1):
- Department of Neurology, Inselspital, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang YZ, Edwards MJ, Rounis E, Bhatia KP, Rothwell JC. Theta burst stimulation of the human motor cortex. Neuron. 2005 Jan 20;45(2):201-6. doi: 10.1016/j.neuron.2004.12.033. PMID 15664172
- [Background] Nyffeler T, Wurtz P, Luscher HR, Hess CW, Senn W, Pflugshaupt T, von Wartburg R, Luthi M, Muri RM. Repetitive TMS over the human oculomotor cortex: comparison of 1-Hz and theta burst stimulation. Neurosci Lett. 2006 Nov 27;409(1):57-60. doi: 10.1016/j.neulet.2006.09.011. Epub 2006 Oct 17. PMID 17049743
- [Result] Cazzoli D, Muri RM, Schumacher R, von Arx S, Chaves S, Gutbrod K, Bohlhalter S, Bauer D, Vanbellingen T, Bertschi M, Kipfer S, Rosenthal CR, Kennard C, Bassetti CL, Nyffeler T. Theta burst stimulation reduces disability during the activities of daily living in spatial neglect. Brain. 2012 Nov;135(Pt 11):3426-39. doi: 10.1093/brain/aws182. Epub 2012 Jul 24. PMID 22831781
- [Result] Marshall L, Helgadottir H, Molle M, Born J. Boosting slow oscillations during sleep potentiates memory. Nature. 2006 Nov 30;444(7119):610-3. doi: 10.1038/nature05278. Epub 2006 Nov 5. PMID 17086200